CLINICAL TRIAL: NCT01340235
Title: Treatment of Dowling Maera Type of Epidermolysis Bullosa Simplex by Oral Erythromycin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Principal Investigator, Del Cont Delphine, Dr Christine CHIAVERINI, Centre Hospitalier Universitaire de Nice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-PP-19
Record Dates: First submitted 2011-04-11; First posted 2011-04-22 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral erythromycin (Experimental): Oral erythromycin
  Interventions: Drug: Oral erythromycin

INTERVENTIONS:
Drug: Oral erythromycin — Severe Dowling Meara EBS patients from 6 months to 8 years old

SUMMARY:
Dowling Meara type of epidermolysis bullosa simplex (EBS-DM) is a rare genodermatosis due to keratin 5 and 14 mutation, characterized by skin fragility and spontaneous or post traumatic blisters. Neonatal period and infancy are critical since this autonomic dominant affection usually improves with age. Cyclins seem to be efficient in some cases of EBS but are prohibited in children younger than 8 years old. Erythromycin can be a good alternative in this population due to its antibacterial and anti-inflammatory potential.

The aim of this study is the evaluation of the efficiency of oral erythromycin to decrease the number of cutaneous blisters in severe EBS-DM patients from 6 months to 8 years old after 3 months of treatment.

Primary end point is the number of patients with decrease of blisters' number of at least 20% after 3 months of treatment by oral erythromycin.

It is a preliminary study on 8 patients. Treatment is oral erythromycin twice a day during 3 months. Follow up for each patient is 5 months. The duration of the study is 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Severe Dowling Meara EBS patients (2 or more new blisters a day)
* signature of informed consent
* Patient of 2 sexes
* Age from 6 months to 8 years. From this age we consider that the patient will less need this treatment or can take cyclines.
* Systematic Obtaining of the consent lit(enlightened) by the relatives(parents) of the child, after information about the objectives and the constraints of the study.
* Agreement of the minor
* Patient member to the Social Security

Exclusion Criteria:

* Patient allergic to the erythromycin
* Patient presenting an intolerance to the fructose, a syndrome of malabsorption some glucose and some galactose or a deficit sucrase-isomaltase
* Renal and\or hepatic Insufficiency
* Patient taking a medicine against indicated or misadvised in association with the erythromycin

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
number of patients with decrease of blisters' number of at least 20% after 3 months of treatment by oral erythromycin | at 3 months of treatment
  Principal end point is evaluated at inclusion and after one month of treatment, 3 months of treatment and 2 months after the end of the treatment

SECONDARY OUTCOMES:
Secondary end points are : effect of 3 months of oral erythromycin on - Global tolerance of treatment. | at 3 months of treatment
  For each patient and globally, the nature, the frequency and the severity of the various unwanted effects will be described on the duration of the study.
Secondary end points are : effect of 3 months of oral erythromycin on - Involved area | at 3 months of treatment
  These criteria will be analyzed in comparison with the values to the inclusion (M0). We shall try to estimate the obstinacy of an effect 2 months after the end of the treatment.
Secondary end points are : effect of 3 months of oral erythromycin on - pruritus, | at 3 months of treatment
  These criteria will be analyzed in comparison with the values to the inclusion (M0). We shall try to estimate the obstinacy of an effect 2 months after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chiaverini, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (4):
- France (4):
  - CHU de Dijon, Dijon
  - Hôpital Saint Eloi, Montpellier
  - CHU de Nice - Hôpital de Cimiez, Nice
  - Hôpital Purpan, Toulouse